CLINICAL TRIAL: NCT05204940
Title: Neurocognitive and Neuroimaging Biomarkers: Predicting Progression Towards Dementia in Patients With Treatment-resistant Late-life Depression (OPTIMUM-Neuro Study)
Brief Title: Longitudinal Observational Biomarker Study
Acronym: OPT-Neuro
Status: Completed | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 080/2017; R01MH114970 (NIH); R01MH114980 (NIH); R01MH114969 (NIH); R01MH114981 (NIH); R01MH114966-01 (NIH)
Record Dates: First submitted 2021-12-24; First posted 2022-01-24 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Depression; Dementia; Mild Cognitive Impairment
MeSH Terms: conditions — Depression; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Investigators will be collecting blood biomarkers as part of their study procedures. These samples will be used to look at other factors that may relate to depression or memory and attention processes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Mechanisms of Late life depression (LLD)-dementia through functional Magnetic Resonance Imaging (fMRI) — Analyzing mechanisms of the LLD-dementia relationship through fMRI acquisitions and analyses, to capture the specific brain networks implicated in executive function and episodic memory decline.
Behavioral: Neuropsychological Data — Neuropsychological Data, including Montreal Cognitive Assessment (MoCA), Wide Range Achievement Test-4 (WRAT-4) Reading subtest, Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) and Delis-Kaplan Executive Function System (D-KEFS) (Color Word Interference, Trail Making and Verbal Fluency).
Behavioral: Clinical Scales — Clinical scales, including the Everyday Cognition Scale (E-Cog), Global Clinical Dementia Rating (CDR), Performance Assessment of Selfcare Skills (PASS)--CIADL (Cognitive Instrumental Activities of Daily Living) Short version, Patient Health Questionnaire (PHQ-9), and Suicide Risk Assessments (Suicide Questions, Baseline Suicidal Ideation, Suicide Intent Scale, Beck Lethality Scale, Decision Outcome Inventory, Columbia-Suicide Severity Rating Scale, and High Suicide Risk Protocol).

SUMMARY:
The purpose of this study is to test whether treatment-resistant late life depression is associated with declines in memory and attention and brain structure and function.

DETAILED DESCRIPTION:
The purpose of this study is to test whether treatment-resistant late life depression is associated with declines in memory and attention and brain structure and function. The study will also test if changes in brain structure and function are associated with decreases in memory. In this study, investigators will conduct a series of assessments/tests, mainly brain imaging and assessments of participant's memory and attention, to better understand how depression is linked to memory and thinking in older persons. Investigators hope that their study will help the scientific community to understand why some people with depressive symptoms that are resistant to treatment in late-life experience declines in their memory and attention and whether effective treatment of such depression reduces that risk. Finally, investigators hope that this study will eventually lead to the development of better treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 60 and older
* Current Major Depressive Disorder (MDD)
* Failure to respond adequately to two or more antidepressant treatment trials of recommended dose and length
* Patient Health Questionnaire-9 (PHQ-9) score of 10 or higher

Exclusion Criteria:

* Dementia
* Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms.
* High risk for suicide and unable to be managed safely in the clinical trial
* Non-correctable, clinically significant sensory impairment interfering with participation
* Unstable medical illness, including delirium, uncontrolled diabetes mellitus, hypertension, hyperlipidemia, or cerebrovascular or cardiovascular risk factors that are not under medical management.
* Moderate to severe substance or alcohol use disorder
* Seizure disorder.
* Parkinson's Disease
* Individuals with any contraindications to MRI

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will recruit 750 patient across all 5 sites who are 60 years or older with Major Depressive Disorder. All participants will be recruited from the OPTIMUM trial (clinicaltrials.gov identifier NCT02960763); all participants who consent and are eligible to participate in OPTIMUM will be invited to participate in this neuroimaging/neurocognitive study. Eligibility bellow will be determined and assessed as per the OPTIMUM clinical trial. In addition, they will have no contra-indications for MRI scanning.
Sampling Method: Non-Probability Sample
Enrollment: 506 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Persistent Depression Leading to Change in Cognition | Baseline, 6-months, 24-months
  To test whether persistent (non-remitting) depression has the ability to change cognition and lead to greater cognitive decline, and greater degradation of neural circuitry

SECONDARY OUTCOMES:
Change in Neural Circuity | Baseline, 6-months, 24-months
  To test whether greater degradation of neural circuitry is associated with greater cognitive decline

CONTACTS AND LOCATIONS:
Overall Officials: Aristotle Voineskos, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (5):
- United States (4):
  - UCLA Late-Life Mood, Stress, and Wellness Research Program, Los Angeles, California
  - Washington University School of Medicine Healthy Mind Lab, St Louis, Missouri
  - Columbia University Adult and Late Life Depression Clinic, New York, New York
  - UPMC Late-Life Depression, Evaluation, Prevention, and Treatment Program, Pittsburgh, Pennsylvania
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
A cleaned, complete, and de-identified copy of the final data set including administrative and technical metadata records will be made available on the National Institute of Mental Health (NIMH) Data Archive and registered at clinicaltrials.gov.
Time Frame: Data will become available after all analyses and initial publication is complete.
Access Criteria: The data will be accessible through the NIMH Data Archive (Collection ID: 2851). Please contact the principal investigators if you have further queries about access criteria.